CLINICAL TRIAL: NCT00811824
Title: Effects of Physical Activity and Dietary Change in Minority Breast Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Heather Greenlee, Assistant Professor, Department of Epidemiology, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: AAAB8839
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: Weight loss; Physical activity; Dietary change
MeSH Terms: conditions — Breast Neoplasms; Weight Loss; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Immediate physical activity and dietary change intervention
  Interventions: Behavioral: Physical activity and dietary change
- 2 (Other): Delayed physical activity and dietary change intervention
  Interventions: Behavioral: Physical activity and dietary change

INTERVENTIONS:
Behavioral: Physical activity and dietary change — 6 months of combined resistance training and aerobic exercise (5 times per week x 30 minutes) plus 6-week nutrition counseling class

SUMMARY:
This study is testing the effects of exercise and dietary change on weight reduction and biological markers associated with breast cancer risk in breast cancer survivors of Hispanic or African descent (n=45). This is a randomized, crossover pilot and feasibility study to test the effects of a 30-minute circuit-based exercise program that combines resistance training with aerobic exercise in conjunction with a low-fat calorie reduced diet. Participants will be randomized to either an immediate 6-months of exercise and dietary change, or a delayed group who will begin their exercise and dietary change program 6-months after the study begins. Participants in the immediate group will be followed for an additional 6-months in order to evaluate adherence to the exercise and dietary change recommendations. Participants in both groups will exercise at a neighborhood Curves® facility at least 5 times per week for six months and will participate in a series of nutrition education classes.

ELIGIBILITY:
Inclusion Criteria:

* 21-70 yrs
* Stage 0-IIIa breast cancer
* No evidence of recurrent/metastatic disease
* Hispanic or African descent (African-American or Caribbean)
* BMI > 25kg/m2
* Sedentary
* Completed surgery, chemotherapy, and radiation therapy ≥ 6 months
* Blood pressure < 140/90
* HgbA1C < 8
* LDL cholesterol < 150
* No uncontrolled comorbidities
* VO2 max normal EKG changes
* Non-smoker

Exclusion Criteria:

* Evidence of recurrent or metastatic breast cancer
* Uncontrolled co-morbid illness including, but not limited to, type I diabetes mellitus, type II diabetes mellitus, hypertension, symptomatic congestive heart failure, unstable angina pectoris, claudication, cardiac arrhythmia; active pulmonary disease; hypercholesterolemia, neurological condition, ischemic heart disease, cardiac disease, kidney disease, respiration problems, asthma, shortness of breath, physical limitations, abnormal thyroid function, active malignancy, except for squamous or basal cell carcinoma of the skin; receiving active chemotherapy or radiotherapy; or psychiatric illness/social situations that would limit compliance with study requirements
* Currently taking Herceptin therapy, or abnormal echo or MUGA post-Herceptin therapy
* Active tobacco use
* Currently active in an exercise and/or dietary change weight loss program
* If a participant develops a breast cancer recurrence or metastasis during the 12-month study period, her participation in the study will be terminated.

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-07; Primary Completion 2009-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Change in weight | 6 months, 12 months
Intervention adherence | 6 months, 12 months

SECONDARY OUTCOMES:
Barriers to participation | 3 months, 6 months, 9 months, 12 months
Predictors of adherence | 3 months, 6 months, 9 months, 12 months
Changes in anthropometric measures | 3 months, 6 months, 9 months, 12 months
Changes in fitness | 3 months, 6 months, 9 months, 12 months
Changes in hormonal biomarkers | 3 months, 6 months, 9 months, 12 months
Changes in metabolic markers | 3 months, 6 months, 9 months, 12 months
Changes in psychological and quality of life measures | 3 months, 6 months, 9 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Heather Greenlee, ND, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Derived] Delgado-Cruzata L, Zhang W, McDonald JA, Tsai WY, Valdovinos C, Falci L, Wang Q, Crew KD, Santella RM, Hershman DL, Greenlee H. Dietary modifications, weight loss, and changes in metabolic markers affect global DNA methylation in Hispanic, African American, and Afro-Caribbean breast cancer survivors. J Nutr. 2015 Apr;145(4):783-90. doi: 10.3945/jn.114.202853. Epub 2015 Feb 4. PMID 25833781